CLINICAL TRIAL: NCT04786171
Title: 4DXV for Targeting in Bronchoscopic Lung Volume Reduction
Brief Title: 4D Medical X-ray Velocimetry for Bronchoscopic Lung Volume Reduction Targeting
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: American Thoracic Society (Other)
Responsible Party: Principal Investigator, Michael Lester, Fellow/Assistant Professor of Pulmonary and Critical Care Medicine, Vanderbilt University Medical Center
Other Study IDs: 12345678910
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Copd; Emphysema; Hyperinflation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 4D X-ray Velocimetry — X-ray velocimetry uses fluoroscopy to quantify local ventilation in the lung.

SUMMARY:
This study will investigate the utility of 4D Medical's X-ray Velocimetry (XV) imaging analysis software for the detection of hyperinflation, and compare endobronchial valve placement outcomes with predictive indices obtained utilizing this technique.

ELIGIBILITY:
Inclusion:

* CT chest and PFTs within the last two years
* Age over 18
* COPD with emphysema
* Global Initiative for Chronic Obstructive Lung Disease (GOLD) 3 - 4 classification OR modified Medical Research Council (mMRC) score of 2 or greater.

Exclusion Criteria:

* Pregnancy
* Presence of an additional pulmonary disease beyond COPD
* Inability to raise arms above 90 degrees as required for fluoroscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with symptomatic emphysema with hyperinflation and no conflating lung diseases or pregnancy.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Ratio of residual volume over functional residual capacity by 4DXV | 6 months
  We will compare an XV hyperinflation index to traditional pulmonary function tests (PFTs) and outcomes
Expiratory Time Constants vs Fissure Completeness | 1 year
  We will examine the correlation between lobar expiratory time constants and fissure completeness by StratX

SECONDARY OUTCOMES:
Improvement in Saint George Respiratory Questionnaire (SGRQ) | 1 year
  We will compare SGRQs pre and post valve placement to hyperinflative indices by 4D XV

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No